CLINICAL TRIAL: NCT01879735
Title: Hepatic Transport of Conjugated Bile Acids in Humans Quantified by 11C-cholylsarcosine PET/CT
Brief Title: Biliary Excretion of Conjugated Bile Acids in Humans Measured by 11C-cholylsarcosine PET/CT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C-CSar humane 244
Record Dates: First submitted 2013-06-11; First posted 2013-06-18 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2014-07

CONDITIONS: Cholestasis; Primary Sclerosing Cholangitis; Primary Biliary Cirrhosis
MeSH Terms: conditions — Cholestasis; Cholangitis, Sclerosing; Liver Cirrhosis, Biliary | interventions — cholylsarcosine; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICG's effect on 11C-CSar transport (Experimental): Examine the effect of ICG on the kinetics of the hepatic transport of 11C-CSar. If no effect is seen on the kinetics, ICG will be used during the "infusion method" experiments.
  Interventions: Drug: 11C-CSar; Drug: ICG
- Infusion method (Experimental): Determine wether bolus or constant infusion of 11C-CSar is optimal for the PET/CT scanning. If ICG does not affect the kinetics of 11C-CSar it will be used during these experiments to calculate hepatic blood flow.
  Interventions: Drug: 11C-CSar; Drug: ICG

INTERVENTIONS:
Drug: 11C-CSar — PET/CT recording with bile acid tracer 11C-cholylsarcosine used to evaluate the transport of bile acids.
  Other Names: 11C-cholylsarcosine
Drug: ICG — Infusion of indocyanine green prior and during the PET/CT scanning with the bile tracer 11C-CSar.
  Other Names: indocyanine green

SUMMARY:
We wish to develop a protocol for PET/CT examination of humans using the bile acid tracer 11C-cholylsarcosine. This is done by a series of PET/CT examinations of healthy humans and patients with cholestatic disorders.

DETAILED DESCRIPTION:
The purpose of the study is the development of PET/CT protocols using 11C-CSar for human use. PET/CT methods developed in the pig studies are translated to studies in healthy humans and patients with cholestatic disorders. Dynamic PET/CT scans of the liver and biliary system are combined with measurements of tracer concentrations in a radial artery and a liver vein and measurements of hepatic blood flow by intravenous infusion of indocyanine green (ICG)/Ficks principle. Kinetic parameters from PET/CT measurements and invasive measurements are compared for validation of the PET estimated parameters and refinement of the PET modeling, if required.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cholestatic disorders and healthy subjects

Exclusion Criteria:

* Body weight above 110 kg (catheterization problematic).
* Diabetes
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Keiding, M.D. D.Sc., Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Nuclear medicine and PET-center, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Derived] Orntoft NW, Munk OL, Frisch K, Ott P, Keiding S, Sorensen M. Hepatobiliary transport kinetics of the conjugated bile acid tracer 11C-CSar quantified in healthy humans and patients by positron emission tomography. J Hepatol. 2017 Aug;67(2):321-327. doi: 10.1016/j.jhep.2017.02.023. Epub 2017 Feb 27. PMID 28249726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 healthy subjects were recruided after they responded to an advertisement in the local newspaper.
  12 patients with varying degree of cholestasis and different underlying diseases were recruided from the Department of hepatology and gastroenterology Aarhus University Hospital.
Groups:
- ICG Infusion: Examine the effect of indocyanine green (ICG) on the hepatic transport of 11C-CSar. Compare the observed kinetics in11C-CSar PET/CT recordings done with and without simultanous infusion of ICG.
- Bolus and Constant Infusion of 11C-CSar: Determine wether bolus or constant infusion of 11C-CSar is optimal for the PET/CT scanning. Two 11C-CSar PET/CT recordings were performed in each subject. One with bolus infusion and one with constant infusion.
Period: Overall Study
Arm/Group | ICG Infusion | Bolus and Constant Infusion of 11C-CSar
Started | 6 | 16
Completed | 6 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ICG's Effect on 11C-CSar Transport: Examine the effect of indocyanine green (ICG) on the rate constants for the hepatic transport of 11C-CSar. Compare the observed kinetics in11C-CSar PET/CT recordings done with and without simultanous infusion of ICG.
- Bolus vs. Constant Infusion: Determine wether bolus or constant infusion of 11C-CSar is optimal for the PET/CT scanning. Two 11C-CSar PET/CT recordings were performed in each subject. One with bolus infusion and one with constant infusion.
- Total: Total of all reporting groups
Arm/Group | ICG's Effect on 11C-CSar Transport | Bolus vs. Constant Infusion | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 12 | 17
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 16 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Whom we Could Quantify Hepatic Transport of 11C-CSar
Time Frame: All measurements are performed in one day.
Measure: Number; unit: percentage of participants
Groups:
- Infusion Method: Determine wether bolus or constant infusion of 11C-CSar is optimal for the PET/CT scanning. Two 11C-CSar PET/CT recordings were performed in each subject. One with bolus infusion and one with constant infusion.
Arm/Group | ICG Infusion | Infusion Method
Number analyzed (Participants) | 6 | 16
percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: Subjects were observed during the PET/CT recordings and for 2 hours after the final PET/CT-recording.
Description: A minor physical examination with blood pressure and puls was performed by a doctor or nurse every 30 minutes for at lest 2 hours after the last PET/CT recording.
Groups:
- ICG's Effect on 11C-CSar Transport: Examine the effect of indocyanine green (ICG) on the hepatic transport of 11C-CSar. Compare the observed kinetics in11C-CSar PET/CT recordings done with and without simultanous infusion of ICG.
Arm/Group | ICG's Effect on 11C-CSar Transport | Bolus vs. Constant Infusion
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 0/6 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes